CLINICAL TRIAL: NCT00346554
Title: To Study the Prevalence of Insomnia in Geriatric COPD Patients Who Are Enrolled in a Pulmonary Rehabilitation Program.
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: 06.01.008
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: COPD; Sleep Disorders
Keywords: COPD; Sleep disorders; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal for COPD patients in pulmonary rehabilitation programs is to improve the quality of life. COPD is known to be worse at night as are other respiratory problems such as CHF. Saturation is known to get worse nocturnally as well. Furthermore, these COPD rehabilitation patients tend to be older and increasing age is associated with an increase in the incidence of sleep disorders. We suspect that there is an increase in the incidence of sleep disorders in COPD patients. We plan to further study these patients using questionnaires. A preliminary study was done, but the results were not comparable to national statistics. We plan to repeat the study, only changing the questions to a format comparable to data from the National Sleep Foundation.

DETAILED DESCRIPTION:
Hackensack University Medical Center Institutional Review Board

PROTOCOL: To study the prevalence of insomnia in geriatric COPD patients who are enrolled in a pulmonary rehabilitation program.

I. OBJECTIVES OF THE STUDY

RATIONALE:

The goal for geriatric patients with COPD and enrolled in pulmonary rehabilitation programs is to improve the quality of life. COPD is known to be worse at night as are other respiratory problems such as CHF. Saturation is known to get worse nocturnally as well. Furthermore, these COPD rehabilitation patients tend to be older, and increasing age is associated with an increase in the incidence of sleep disorders. We suspect that there is an increase in the incidence of difficulty initiating and maintaining sleep in COPD patients. A preliminary study was done by the chest medicine specialist in our group, but the results were not comparable to national statistics and were inconclusive. We plan to further evaluate the geriatric COPD patients in pulmonary rehabilitation with initial screening questionnaire and diagnostic screening questionnaires (MMSE, Beck's Anxiety Inventory, Beck's Depression Inventory, and Epworth Sleepiness Scale).

GOALS:

* To determine the incidence and prevalence of insomnia (difficulty initiating sleep (DIS), and/or difficulty maintaining sleep (DMS) in the geriatric population with COPD in a rehabilitation program.
* To determine how many of these patients suffer from anxiety and/or depression.

HYPOTHESIS:

The incidence of insomnia (DIS and/or DMS), along with anxiety/depression is more prevalent in geriatric patients with COPD.

II. BACKGROUND MATERIAL According to the American Academy of Sleep Medicine (AASM), over a six-month period, 20 million Americans complained of insomnia.

COPD patients tend to have decreased total sleep time (32% reported total sleep time less than 6 hours). According to previous studies conducted, the following was reported:

* 15% reported to have insomnia;
* 28% reported poor quality sleep due to anxiety and/or depression;
* 12% reported > 3 awakenings due to unknown origin.

RESULTS OF PILOT:

In the pilot study, a preliminary general (initial) questionnaire was used and will continue to be used as a tool for general screening purposes. And diagnostic questionnaires will be used, which are the following:

* Beck's Anxiety Inventory
* Beck's Depression Inventory
* Epworth Sleepiness Scale
* MMSE

III. DRUG INFORMATION

No drugs are used in this study protocol.

IV. INCLUSIONARY CRITERIA

Geriatric patients with COPD enrolled in the rehabilitation program with FEV1<60%.

V. EXCLUSIONARY CRITERIA

Geriatric patients without a clear diagnosis of COPD. Geriatric patients whose FEV1>60%. Geriatric patients who are unable to answer the questionnaire.

VI. RECRUITMENT PROCEDURES

Geriatric patients in the HUMC pulmonary rehabilitation program who consent to answer the questionnaire and with an FEV1<60% will be enrolled.

VII. METHODOLOGY

Screening: Charts will be reviewed to see which patients meet the criteria of the study.

Informed Consent: If the patient is eligible for diagnostic screening, then an informed consent will be taken.

Randomization: None

Baseline evaluation: Geriatric patients will be asked the questions in the questionnaire.

Follow-up: If insomnia is found, patient will be referred for further treatment.

Withdrawal and Termination: The patient is unable to complete the questionnaire.

VIII. DISCOMFORT AND RISKS

No direct risks to the patient. Failure to follow-up in the clinic if indicated could be problematic.

IX. BENEFITS

Recognition and treatment of sleep problems in this group of patients will add to our understanding of problems in COPD.

X. CRITERIA FOR EVALUATING RESPONSE

No response anticipated from the study protocol.

XI. CONFIDENTIALITY

All results will be kept confidential. Data will only be used by the investigators. Data can be reviewed by the IRB at any time. HIPPA forms will be used for the patient's permission.

XII. PRIMARY INVESTIGATOR

Hormoz Ashtyani, M.D.

CO PRIMARY INVESTIGATOR

Susan Zafarlotfi Ph.D

GERIATRIC MEDICINE SPECIALIST

Knight R. Steel, M.D.

RESEARCH COORDINATOR

Mohammad Quadri, M.D. (MBA) RPSGT

ELIGIBILITY:
Inclusion Criteria:

* COPD
* rehabilitation program
* FEV1<60%

Exclusion Criteria:

* FEV1>60%

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Greitric COPD patients who are enrolled in Pulmonary Rehabilitation at HUMC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hormoz Ashtyani, MD, Principal Investigator — Hackensack Meridian Health; Susan Zafarlotfi, Ph.D, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center - Pulmonary Rehabilitation, Hackensack, New Jersey, United States